CLINICAL TRIAL: NCT05808842
Title: Evaluation of the UltraClear Laser Workstation for the Treatment of Facial and Neck Rejuvenation and Skin Resurfacing Augmented With Mesenchymal Stem Cell Extract
Brief Title: Laser Treatment for Facial and Neck Rejuvenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Acclaro Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UC 16-2022
Record Dates: First submitted 2023-03-20; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Face Rejuvenation; Neck Rejuvenation
Keywords: Wrinkles; Fine Lines; Sun Spots; Laxity; Facial Laxity
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to have one of two post-laser skincare regimens which will be applied to the face and neck following laser treatment.
Who Masked: Investigator
Masking Description: The blinded investigator will complete the - Fitzpatrick-Goldman Classification of Wrinkling and Degree of Elastosis Scale of face and neck, the Scientific Assessment Scale of Skin Quality (SASSQ) to grade the subject's skin quality of face and neck, the Classification of Facial Wrinkles Assessment and the Blinded Investigator Neck Skin Crepiness/Laxity Grading Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A CeraVe (Active Comparator): Subjects will be given a skincare regimen consisting of CeraVe products to be applied to the face and neck following laser treatment.
  Interventions: Other: CeraVe
- Group B Calecim (Sham Comparator): Subjects will be given a skincare regimen consisting of CeraVe products and Calecim products to be applied to the face and neck following laser treatment.
  Interventions: Other: CeraVe and Calecim

INTERVENTIONS:
Other: CeraVe — * CeraVe gentle facial cleanser (CeraVe; New York, NY) to be used morning and evening
  * CeraVe lotion (CeraVe; New York, NY) to be used morning and evening, reapply as needed for dry skin
  * A mineral CeraVe sunscreen (CeraVe; New York, NY) to be applied in the morning and reapplied every 2 hours if going outside
  Arms: Group A CeraVe
Other: CeraVe and Calecim — * CeraVe gentle facial cleanser (CeraVe; New York, NY) to be used morning and evening
  * Calecim® Professional Serum (CellResearch Corporation; Singapore) to be used morning and evening
  * Calecim® Restorative Hydration Cream (CellResearch Corporation; Singapore) to be used morning and evening, reapply as needed for dry skin
  * A mineral CeraVe sunscreen (CeraVe; New York, NY) to be applied in the morning and reapplied every 2 hours if going outside
  Arms: Group B Calecim

SUMMARY:
To assess the efficacy, safety, and patient satisfaction associated with the treatment of the face and neck with the 2,910nm mid-infrared UltraClear Laser System using both superficial epidermal ablation and deep ablative and coagulative capabilities in the dermis for rejuvenation of photodamaged skin. Additionally, this study will assess the additive value of a post-treatment skincare regimen consisting of a serum and cream containing red deer umbilical cord lining mesenchymal stem cell conditioned media for faster healing and more robust rejuvenation.

DETAILED DESCRIPTION:
Subjects will be treated with the UltraClear 2,910nm mid-infrared laser using both superficial epidermal ablation and deep ablative and coagulative capabilities in the dermis for rejuvenation of photodamaged skin of the face and neck. Subjects will be randomized to have one of two post-laser skincare regimens which will be applied to the face and neck following laser treatment.

All subjects will receive three (3) laser treatments to the face and neck using the UltraClear 2,910nm mid-infrared laser, performed 5 weeks ± 7 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18 to 75 years
* Fitzpatrick skin types I-V
* Subjects in good general health based on investigator's judgment and medical history
* Must be willing to give and sign an informed consent form and photographic release form
* Willingness to have examinations of face and neck and digital photographs performed of the face and neck
* Physician evaluator classifying the subject as moderate to severe (Class II-III, Score 4-9) on the Fitzpatrick-Goldman Classification of Wrinkling and Degree of Elastosis Scale for the face and neck.
* The subject must be planning to undergo fractional ablative laser resurfacing to the face and neck and be willing to comply with study protocol and complete the entire course of the study.
* Subjects using any treatment skincare products (per investigator discretion) must discontinue use of these products before the start of participating in this clinical study and for the duration of the study.
* Male subjects with facial hair must be willing to shave the morning of the procedure.
* Must be willing to maintain usual sun exposure
* Subject agrees to avoid tanning or use of sunless tanner during the entire course of the study
* Negative urine pregnancy test result at the time of study entry (if applicable)
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

  1. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
  2. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.
* Must be willing to comply with study treatments and complete the entire course of the study

Exclusion Criteria:

* Energy-based device (i.e., radiofrequency device treatments, microfocused ultrasound device or other ultrasound-based device treatments, laser and light-based device treatments, microneedling) treatment in the treatment area in the last 6 months
* Chemical peel or microdermabrasion of the face within 30 days prior to enrollment in the study
* Surgery (i.e., face lift, eyebrow lift, neck lift or lower rhytidectomy, liposuction to the neck and/or submentum, etc.) during the 12-month period before study treatment
* Any investigational treatment for improvement of skin quality and/or photodamage of facial skin during the 12-month period before the study treatment
* Recent use of topical tretinoin, adapalene, tazarotene, hydroquinone, imiquimod, 5-fluorouracil, ingenol mebutate, concentrated hydrogen peroxide, diclofenac, or photodynamic therapy (PDT) to the face within the previous 4 weeks
* Subjects must not currently be taking isotretinoin (Accutane).
* Creams/cosmeceuticals and/or home therapies to prevent or treat photodamage, uneven skin pigmentation, excessive erythema (redness), fine lines/wrinkles, skin laxity and/or pore size during the 4-week period before study treatment
* Subjects with scarring in the treatment areas
* Subjects with tattoos or permanent implants in the treatment areas
* Subjects with a significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study
* Subjects with a history of or presence of any skin condition/disease (including but not limited to any visible rash, atopic dermatitis, psoriasis, actinic keratoses, keratinocyte carcinoma, melanoma, etc.) in the treatment area that might interfere with the diagnosis or evaluation of study parameters
* Skin with open wounds, excessively sensitive skin, neurotic excoriations, dermatitis or inflammatory rosacea in the treatment area
* History of keloid or hypertrophic scarring
* Subjects with an active bacterial, viral, or fungal infection of the treatment areas or systemic infection
* Subjects who spray tanned or used sunless tanners in the treatment areas four (4) weeks prior to study treatment
* History of lidocaine and/or tetracaine sensitivity deemed by the investigator to preclude the subject from enrolling into the study
* Individuals with known allergies or sensitivities to any of the ingredients of any topical products being used in this study
* Subjects must not have a compromised ability for wound healing, such as: malnutrition, steroid use, history of collagen vascular disease (e.g., lupus, scleroderma), atopic dermatitis, or immunologic abnormalities such as vitiligo.
* Subjects planning any cosmetic procedure to the treatment areas during the study period, other than the treatment that will be performed by the investigator
* Presence of incompletely healed wound(s) in the treatment area
* Subjects who are on an immunosuppressant or have an autoimmune condition
* Female subjects who are pregnant, planning a pregnancy, or breast feeding during the study
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-03 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Fitzpatrick-Goldman Classification of Wrinkling and Degree of Elastosis Scale to assess change (blinded investigator) | Baseline, Day 60, Day 250
  Fitzpatrick-Goldman Classification of Wrinkling and Degree of Elastosis Scale - FACE TO BE COMPLETED BY BLINDED INVESTIGATOR
  Class: Wrinkling Score Degree of Elastosis
  I Fine Wrinkles 1 -3 Mild
  II Fine to Moderate 4 -6 Moderate
  III Fine to Deep 7 -9 Severe
Scientific Assessment Scale of Skin Quality to assess change (SASSQ) (blinded investigator) | Baseline, Day 160, Day 250
  SCIENTIFIC ASSESSMENT SCALE OF SKIN QUALITY (SASSQ)
  Elasticity:
  0-None 1-Mild 2-Moderate 3-Severe 4-Very Severe
  Wrinkles:
  0-None 1-Mild 2-Moderate 3-Severe 4-Very Severe
  Skin Surface Roughness:
  0-None 1-Mild 2-Moderate 3-Severe 4-Very Severe
  Pigmentation:
  0-None 1-Mild 2-Moderate 3-Severe 4-Very Severe
  Erythema:
  0-None 1-Mild 2-Moderate 3-Severe 4-Very Severe
  Pore Size:
  0-None 1-Mild 2-Moderate 3-Severe 4-Very Severe
Classification of Facial Wrinkles Assessment to assess change (blinded investigator) | Baseline, Day 160, Day 250
  Classification of Facial Wrinkles Assessment:
  Preauricular Lines:
  0-None 1-Very Mild 2-Mild 3-Moderate 4-Severe 5-Extreme
  Cheek Folds:
  0-None 1-Very Mild 2-Mild 3-Moderate 4-Severe 5-Extreme
  Upper Lip Lines:
  0-None 1-Very Mild 2-Mild 3-Moderate 4-Severe 5-Extreme
Neck Skin Crepiness/Laxity Grading Scale to assess change (blinded investigator) | Baseline, Day 160, Day 250
  Neck Skin Crepiness/Laxity Grading Scale:
  Score Classification Description 0 None No Loose Skin
  1. Mild Mildly Loose Skin
  2. Moderate Moderately Loose Skin
  3. Severe Very Loose Skin
  4. Extreme Prominent redundancy of loose skin
Visia Skin Analysis to assess change | Baseline, Day 160, Day 250
  Visia Skin Analysis (insert percentage 1 - 100%)
  Description: Percentage:
  Brown Spots Pores Spots Porphyrin Red Areas Texture UV Spots Wrinkles
Physician Global Aesthetic Improvement Scale to assess change (PGAIS) (blinded investigator) | Day 160, Day 250
  Physician Global Aesthetic Improvement Scale Assessment (PGAIS) Rating Description
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re- treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.
  Scores (write a number under each treated area or circle "Not Treated")
  FACE NECK
  not treated not treated
Percent Improvement Evaluation to assess change | Day 160, Day 250
  Percent Improvement Evaluation:
  Degree of improvement from clinical evaluation, compare to baseline, using a 1-10 scale.
  1 (0-10%) 2 (10-20%) 3 (20-30%) 4(30-40%) 5 (40-50%)
  6 (50-60%) 7 (60-70%) 8 (70-80%) 9 (80-90%) 10 (90-100%)

SECONDARY OUTCOMES:
Evaluation of side effects and adverse events by Investigator to assess change | Baseline, Day 35, Day 70, Day 160, Day 250
  Evaluation of Side Effects and Adverse Events:
  Rating Description 0 NONE: Normal
  1. TRACE: Barely visible and localized
  2. MILD: Somewhat visible and diffuse
  3. MODERATE: Visible and diffuse
  4. SEVERE: Extremely visible and dense
  SCORES (write number under each treated area or check "Not Treated")
  Erythema:
  FACE NECK
  Edema:
  FACE NECK
  Hyperpigmentation:
  FACE NECK
  Blistering:
  FACE NECK
  Burn:
  FACE NECK
  Skin Crusting:
  FACE NECK
Comfort Level Visual Analog Scale post laser procedure to assess change (completed by subject) | Baseline, Day 35, Day 70
  Comfort Level Visual Analog Scale post laser procedure (circle one)
  Face:
  No Pain Moderate Pain Worst Pain
  0 1 2 3 4 5 6 7 8 9 10
  Neck:
  No Pain Moderate Pain Worst Pain
  0 1 2 3 4 5 6 7 8 9 10
Subject Global Aesthetic Improvement Scale to assess change (SGAIS) | Day 160, Day 250
  Subject Global Aesthetic Improvement Scale Assessment (SGAIS)
  Rating Description
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re- treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.
  Scores (write a number under each treated area or circle Not Treated)
  FACE NECK
  not treated not treated
Subject Satisfaction Questionnaire to assess change | Day 160, Day 250
  Subject Satisfaction Questionnaire
  How would you rate your satisfaction of each treated area? Non-treated areas will be checked as "Not Treated" for you.
  Rating Description 0 Not satisfied
  1. Somewhat satisfied
  2. Satisfied
  3. Very satisfied
  4. Extremely Satisfied
  Scores (write a number to rate each treated area) FACE NECK
  not treated not treated

IPD SHARING:
Plan to Share IPD: Undecided